CLINICAL TRIAL: NCT02994212
Title: Reduced Frequency of Visits in the Treatment of Uncomplicated Severe Acute Malnutrition: Evaluation of Operational Feasibility and Safety
Brief Title: Reduced Visit Frequency in the Treatment of Uncomplicated Severe Acute Malnutrition: Evaluation of Operational Feasibility and Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Epicentre (Other)
Collaborators: Médecins Sans Frontières, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 821414-1
Record Dates: First submitted 2016-12-13; First posted 2016-12-15 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Severe Acute Malnutrition
MeSH Terms: conditions — Severe Acute Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention group (Experimental): 115 children eligible for the outpatient treatment of SAM were provided a monthly ration of RUTF. Anthropometric measurements were taken on a weekly basis for 4 weeks to monitor treatment response.
  Interventions: Dietary Supplement: Monthly distribution of RUTF

INTERVENTIONS:
Dietary Supplement: Monthly distribution of RUTF — 115 children eligible for the outpatient treatment of SAM were provided a monthly ration of RUTF.

SUMMARY:
Community-based management of severe acute malnutrition (SAM) has been shown to be safe and cost-effective, but program coverage remains low. New treatment models that maintain high levels of clinical effectiveness but allow for increased coverage are still needed. A reduced schedule of follow-up, in which children receive clinical follow-up and therapeutic foods on a monthly rather than weekly or biweekly basis, may be one alternative. This study aims to describe the safety and feasibility of a monthly distribution of ready-to-use therapeutic food in the treatment of uncomplicated SAM, in terms of clinical response to treatment and household ready-to-use therapeutic food (RUTF) utilization. This is a non-randomized pilot intervention study in which 115 children eligible for the outpatient treatment of SAM were provided a monthly ration of RUTF. Anthropometric measurements were taken on a weekly basis for 4 weeks to monitor treatment response defined as weight gain, (mid-upper arm circumference) MUAC gain, weight loss > 5%, and the development of edema. Unannounced household spot checks were conducted over 4 weeks to assess household utilization of RUTF and storage practices.

ELIGIBILITY:
Inclusion Criteria:

* a) being eligible for new admission to treatment of uncomplicated SAM
* b) being resident within 15 km of the study health center

Exclusion Criteria:

* previously default from previous SAM treatment (e.g. missed 2 consecutive weekly visits)
* considered a relapse case (e.g. re-admitted within three months of previous discharge)

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 115 (Actual)
Dates: Start 2014-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
weight gain | 4 weeks
  grams/kilograms/day gained
mid-upper arm circumference gain (mm/day) | 4 weeks
  millimeters gained per day
weight loss > 5% | 4 weeks
development of edema | 4 weeks

SECONDARY OUTCOMES:
correct utilization of RUTF | 4 weeks
  > 2 sachets deviance between available and expected RUTF stocks at unannounced household visits

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Isanaka, ScD, Principal Investigator — Epicentre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Isanaka S, Kodish SR, Berthe F, Alley I, Nackers F, Hanson KE, Grais RF. Outpatient treatment of severe acute malnutrition: response to treatment with a reduced schedule of therapeutic food distribution. Am J Clin Nutr. 2017 May;105(5):1191-1197. doi: 10.3945/ajcn.116.148064. Epub 2017 Apr 12. PMID 28404577